CLINICAL TRIAL: NCT02281084
Title: A Phase 2, International, Multicenter, Randomized, Open-label, Parallel Group to Evaluate the Efficacy and Safety of Cc-486 (Oral Azacitidine) Alone in Combination With Durvalumab (MEDI4736) in Subjects With Myelodysplastic Syndromes Who Fail to Achieve an Objective Response to Treatment With Azacitidine for Injection or Decitabine
Brief Title: Safety and Efficacy Study of CC-486 in Subjects With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-486-MDS-006; 2014-002675-29 (EudraCT Number)
Expanded Access: NCT03723135 (Approved for marketing)
Record Dates: First submitted 2014-10-21; First posted 2014-11-03 (Estimated); Results first posted 2020-07-08 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Myelodysplastic Syndromes
Keywords: Keywords provided by Celgene:; myelodysplastic syndromes; MDS; azacitidine; oral azacitidine (CC-486); decitabine; intermediate-1; intermediate-2 and high risk myelodysplastic syndromes (MDS); proliferative chronic myelomonocytic leukemia (CMML); Chronic; iHMA (injectable hypomethylating agents); PD-L1
MeSH Terms: conditions — Myelodysplastic Syndromes; Bronchiolitis Obliterans Syndrome | interventions — Azacitidine; cc-486; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monotherapy: Oral Azacitidine (Experimental): Oral azacitidine (AZA) 100 mg, 150 mg, or 200 mg tablets twice daily (BID) on days 1 to 21 of each 28-day treatment cycle. Participants continued to receive their assigned study treatment unless disease progression, unacceptable toxicity, lost to follow-up or withdrawal by participant occurred.
  Interventions: Drug: Oral Azacitidine
- Combination Therapy: Oral Azacitidine and Durvalumab (Experimental): Oral Azacitidine 100 mg oral azacitidine tablets BID on days 1 to 14 or days 1 to 21 of each 28-day treatment cycle and durvalumab 1500 mg by intravenous (IV) infusion on day 1 of each 28-day treatment cycle; participants continued to receive their assigned study treatment unless disease progression, unacceptable toxicity, lost to follow-up or withdrawal by participant occurred.
  Interventions: Drug: Oral Azacitidine; Drug: Durvalumab

INTERVENTIONS:
Drug: Oral Azacitidine — Oral azacitidine (AZA) 100 mg, 150 mg, or 200 mg tablets twice daily (BID) on days 1 to 21 of each 28-day treatment cycle. Participants continued to receive their assigned study treatment unless disease progression, unacceptable toxicity, lost to follow-up or withdrawal by participant occurred.
  Other Names: CC-486
Drug: Durvalumab — Durvalumab 1500 mg by IV infusion on Day 1 of each 28 day treatment cycle.
  Other Names: Imfinzi; MEDI4736
  Arms: Combination Therapy: Oral Azacitidine and Durvalumab

SUMMARY:
Evaluate the safety and efficacy of oral azacitidne (CC-486) twice daily (BID) in subjects with myelodysplastic syndromes who failed to achieve an objective response post injectable hypomethylating agent (iHMA) treatment

Reason for removing the combination arm: Due to difficulties with dose-finding, the durvalumab plus CC-486 combination arm was closed to enrollment.

Extension:

An Extension Phase (EP) has been added to allow subjects who are currently receiving oral azacitidine BID and who are demonstrating clinical benefit as assessed by the Investigator, to continue receiving oral azacitidine until the subject meets the criteria for study discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 18 years of age at the time of signing the informed consent document
2. Documented diagnosis of MYELODYSPLASTIC SYNDROMES (MDS), classified according to FRENCH-AMERICAN BRITISH (FAB) classification criteria
3. Adequate course of treatment with an injectable hypomethylating agent (azacitidine for injection or decitabine) as the last therapeutic intervention for MDS prior to beginning screening for this study. Adequate is defined as:

   * having received at least 6 consecutive 4-week treatment cycles with azacitidine for injection, or
   * having received at least 4 consecutive 6-week treatment cycles with decitabine (3-day regimen) or at least 6 consecutive 4-week treatment cycles with decitabine (5-day regimen), or
   * having demonstrated inability to tolerate treatment with an injectable hypomethylating agent because of unacceptable drug-related toxicity after at least 3 months of attempted treatment: Three 28-day cycles of azacitidine for injection or decitabine 5-day regimen; two 42-day cycles of decitabine 3-day regimen.
4. Documented disease progression or stable disease as best response to treatment (or attempted treatment) with azacitidine for injection or decitabine. Those achieving an objective response to treatment regimen with an injectable hypomethylating agent (HMA) are excluded from participation in this study.

   Definitions of disease progression are modified from INTERNATIONAL WORKING GROUP (IWG) 2006 criteria and include:

   - Pre-injectable hypomethylating agent baseline bone marrow myeloblasts:
   1. Less than 5%: ≥ 100% increase to ≥ 8% blasts
   2. ≥ 5%: ≥ 50% increase to ≥ 10% blasts Note: ≥ 30% blasts is considered acute myeloid leukemia (AML )per FAB classification. Subjects known to have ≥ 30% blasts are not eligible for inclusion in this study.recognizing eastern cooperative oncology group) limitations of blast cell quantification, Protocol will allow subjects with pre-enrollment bone marrow blast counts up to 33% on the screening bone marrow examination to be considered for inclusion. Assessment may be made according to local bone marrow examination to facilitate enrollment of eligible subjects into the treatment phase of the study.

      - Any clinical worsening from pre-injectable hypomethylating agents (HMA) baseline condition, including:

   <!-- -->

   1. sustained clinically-significant worsening (investigator's assessment) from baseline granulocyte, platelet, or hemoglobin values (≥ 2 values, separated by ≥ 2 weeks) - worsening granulocytes should be ≥ 50% decrease from pre-injectable HMA baseline value - worsening platelets should be ≥ 50% decrease from pre-injectable HMA baseline value (untransfused)

      * worsening hemoglobin should be ≥ 1.5 g/dL decrease from preinjectable HMA baseline value in subjects not receiving RBC transfusions
   2. meaningful worsening in RBC or platelet transfusion requirement

      Definition of stable disease is based on modified IWG 2006 criteria:
      * Failure to achieve any objective response (CR - complete remission, PR - partial remissino, mCR - marrow complete remission, or HI - hematologic improvement), but no evidence of disease progression within the 8 weeks leading to the subject's first dose of investigational product (IP), Cycle 1, Day 1
5. Have the last dose of the prior treatment regimen injectable HMA - (azacitidine for injection or decitabine) not more than 16 weeks prior to screening for this study (date of informed consent signature).
6. No less than 3 weeks between the last dose of the prior treatment regimen injectable HMA - (azacitidine for injection or decitabine) and the planned date of first dose of IP (
7. Have an eastern cooperative oncology group (ECOG) performance status of 0, 1, or 2
8. Females subjects of childbearing potential (FCBP)1 may participate, providing they meet the following conditions:

   1. Have two negative pregnancy tests as verified by the investigator prior to starting any IP therapy: serum pregnancy test at screening and negative serum or urine pregnancy test (investigator's discretion) within 72 hours prior to starting treatment with IP (Cycle 1, Day 1). They must agree to ongoing pregnancy testing during the course of the study (before beginning each subsequent cycle of treatment), and after the last dose of any IP. This applies even if the subject practices complete abstinence2 from heterosexual contact.
   2. Agree to practice true abstinence2 (which must be reviewed on a monthly basis and source documented) or agree to the use of highly effective methods of contraception from 28 days prior to starting azacitidine, and must agree to continue using such precautions while taking azacitidine (including dose interruptions) and for up to 90 days after the last dose of azacitidine. Cessation of contraception after this point should be discussed with a responsible physician
   3. Agree to abstain from breastfeeding during study participation and for at least 90 days after the last dose of IP.

Note that the screening serum pregnancy test can also be used as the test prior to starting IP if it is performed within the 72-hour timeframe.

9. Male subjects must:

1. Male subjects must:

   1. Either practice true abstinence2 from heterosexual contact (which must be reviewed on a monthly basis) or agree to avoid fathering a child, to use highly effective methods of contraception, male condom plus spermicide during sexual contact with a pregnant female or a female of child bearing potential (even if he has undergone a successful vasectomy) from starting dose of IP (Cycle 1 Day 1), including dose interruptions through 90 days after receipt of the last dose of azacitidine.
2. Refrain from semen or sperm donation while taking IP and for at least 90 days after the last dose of IP.

   10. Understand and voluntarily sign an informed consent document prior to any study-related assessments or procedures conducted.

   11. Be able to adhere to the study visit schedule and other protocol requirements.

   12. Understand and voluntarily sign a biomarker-specific component of the informed consent document prior to any study-related procedures conducted.

Extension Phase

At the Investigator's discretion and following confirmation of eligibility criteria below, subjects can enter the Extension Phase (EP):

* Subjects who have signed the informed consent for the EP of the study;
* Subjects receiving oral azacitidine and continuing in the treatment phase demonstrating clinical benefit as assessed by the Investigator are eligible to receive oral azacitidine in the EP;
* Subjects who do not meet any of the criteria for study discontinuation

Exclusion Criteria:

1. Rapidly-progressing MDS defined as:

   1. Known clinically-significant doubling in marrow or per IP peripheral blood blast percentage (to ≥ 20%) in the 8-week period leading to the first dose of IP (Cycle 1, Day 1)
   2. ≥100% increase in WBC count (myeloid cell line and monocyte series) within the 8-week period leading to Cycle 1, Day 1
2. AML - FAB (FRENCH-AMERICAN-BRITISH) classification: ≥ 30% blasts in bone marrow). Subjects known to have ≥ 30% blasts are not eligible for inclusion in this study. Recognizing limitations of blast cell quantification, this protocol will allow subjects with pre-enrollment (screening/baseline) bone marrow blast counts up to 33% to be considered for inclusion.
3. Prior allogeneic stem cell transplant
4. Prior exposure to the investigational oral formulation of decitabine, or other oral azacitidine derivative at any time in the subject's prior history
5. Prior or ongoing response (IWG 2006: HI, PR, CR, or marrow CR) to treatment with azacitidine for injection or decitabine, at any time in the subject's prior history, which includes relapsed disease
6. Ongoing medically significant adverse events from previous treatment, regardless of the time period
7. Use of any of the following within 28 days prior to the first dose of IP:

   1. thrombopoiesis-stimulating agents ([TSAs]; eg, Romiplostim, Eltrombopag, Interleukin-11)
   2. ESAs (Erythropoiesis stimulating agent) and other RBC hematopoietic growth factors (eg, interleukin-3)
   3. hydroxyurea
8. Concurrent use of corticosteroids unless the subject is on a stable or decreasing dose for ≥ 1 week prior to enrollment for medical conditions other than MDS
9. History of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis), celiac disease (ie, sprue), prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with the absorption, distribution, metabolism or excretion of the IP and/or predispose the subject to an increased risk of gastrointestinal toxicity
10. Prior history of malignancies, other than MDS, unless the subject has been free of the disease for ≥ 3 years. However, subjects with the following history/concurrent conditions are allowed:

    1. Basal or squamous cell carcinoma of the skin
    2. Carcinoma in situ of the cervix
    3. Carcinoma in situ of the breast
    4. Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, nodes, metastasis [TNM] clinical staging system)
11. Significant active cardiac disease within the previous 6 months, including:

    1. New York Heart Association (NYHA) class IV congestive heart failure;
    2. Unstable angina or angina requiring surgical or medical intervention; and/or
    3. Myocardial infarction
12. Uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment)
13. Known Human Immunodeficiency Virus (HIV) or Hepatitis C (HCV) infection, or evidence of active Hepatitis B Virus (HBV) infection
14. Any of the following laboratory abnormalities:

    1. Serum Aspartate transaminase / Serum glutamic oxaloacetic transaminase (AST/SGOT) Alanine aminotransaminase / Serum glutamic pyruvate transaminase (ALT/SGPT) > 2.5 x ULN (upper limit of normal)
    2. Serum total bilirubin > 1.5 x upper limit of normal (ULN). Higher levels are acceptable if these can be attributed to active red blood cell precursor destruction within the bone marrow (ie, ineffective erythropoiesis). Subjects are excluded if there is evidence of autoimmune hemolytic anemia manifested as a corrected reticulocyte count of > 2% with either a positive Coombs' test or over 50% of indirect bilirubin
    3. Serum creatinine > 2.5 x ULN (upper limit of normal)
    4. Absolute WBC (white blood cell) count ≥ 20 x 109/L
15. Known or suspected hypersensitivity to azacitidine, mannitol, its constituents, or to any other humanized monoclonal antibody
16. Pregnant, planning to become pregnant starting from 28 days prior to receiving CC-486 throughout your participation in the study, and for at least 90 days following your last dose of study treatment, or breast-feeding females
17. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
18. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
19. Any condition that confounds the ability to interpret data from the study, including known or suspected conditions other than MDS, associated with anemia
20. Having received any prior MAb (monoclonal antibodies) against CTLA-4 (cytotoxic T lymphocyte-associated antigen), PD-1, or PD-L1 or having received other investigational monoclonalantibodies (MAbs) within 6 months
21. Clinical evidence of central nervous system (CNS) or pulmonary leukostasis, or CNS leukemia
22. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis, Crohn's disease], diverticulitis with the exception of a prior episode that has resolved or diverticulosis, celiac disease, irritable bowel disease, or other serious gastrointestinal chronic conditions associated with diarrhea; systemic lupus erythematosus; Wegener's syndrome [granulomatosis with polyangiitis]; myasthenia gravis; Graves' disease; rheumatoid arthritis; hypophysitis, uveitis; etc) within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:

    1. Subjects with vitiligo or alopecia;
    2. Subjects with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement for ≥ 3 months; or
    3. Subjects with psoriasis not requiring systemic treatment
23. History of primary immunodeficiency
24. Active myeloproliferative neoplasms (MPN) and chronic myelomonocytic leukemia (CMML)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-07-06 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2023-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (89):
- United States (23):
  - Local Institution - 113, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - University of Miami Miller School of Medicine, Miami, Florida
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Local Institution - 104, Tampa, Florida
  - Local Institution - 111, Chicago, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Local Institution - 109, Harvey, Illinois
  - Local Institution - 116, Iowa City, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Local Institution - 103, Louisville, Kentucky
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Local Institution - 102, Hackensack, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Local Institution - 101, New York, New York
  - Local Institution - 110, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Hillman Cancer Institute at UPMC, Pittsburgh, Pennsylvania
  - University of Texas- MD Anderson, Houston, Texas
  - Cancer Care Centers of South Texas - HOAST, San Antonio, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (9):
  - Westmead Hospital, Westmead, New South Wales
  - Local Institution - 401, Adelaide, South Australia
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Local Institution - 400, Clayton, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - Local Institution - 405, Malvern, Victoria
  - Royal Brisbane and Women's Hospital, Herston
  - Royal Perth Hospital, Perth
- Belgium (7):
  - Hopital Erasme, Brussels
  - Local Institution - 802, Brussels
  - Local Institution - 801, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Centre Hospitalier Universitaire de Liege, Liège
  - Local Institution - 800, Liège
  - Clinique Saint-Pierre, Ottignies
- Local Institution - UNK-004, Hamilton, Ontario, Canada
- France (4):
  - Institut Paoli Calmettes, Marseille
  - Hopital Saint-Louis, Paris
  - Local Institution - 201, Paris
  - CHU Purpan, Toulouse
- Germany (8):
  - Local Institution - 500, Dresden
  - Universitatsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Local Institution - 502, Düsseldorf
  - Marien Hospital, Düsseldorf
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Universitatsklinikum Halle Saale, Halle
  - Universitatsklinikum Leipzig, Leipzig
  - Medizinische Klinik III Klinikum der Universität München-Großhadern, München
- Italy (7):
  - Azienda Ospedaliera Santi Antonio Biagio E Cesare Arrigo, Allessandria
  - Azienda Ospedaliera Universitaria Policlinico Sant Orsola Malpighi, Bologna
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Local Institution - 601, Florence
  - Ospedale San Raffaele S.r.l., Milan
  - Azienda Ospedaliera Sant Andrea, Roma
  - Local Institution - 603, Roma
- Poland (4):
  - Zaklad Opieki Zdrowotnej MSW z Warminsko-Mazurskim Centrum Onkologii, Olsztyn
  - Local Institution - 900, Warsaw
  - MTZ Clinical Research Sp. z o.o., Warsaw
  - Uniwersytecki Szpital Kliniczny, Wroclaw
- Spain (15):
  - Institut Calatà d'Oncologia, L'Hospitalet, Barcelona
  - Local Institution - 306, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Virgenes de las Nieves, Granada
  - Local Institution - 300, Granada
  - Hospital General Gregorio Maranon, Madrid
  - Local Institution - 307, Madrid
  - Hospital Universitario Virgen De La Victoria, Málaga
  - Hospital Central de Asturias, Oviedo
  - Local Institution - 303, Oviedo
  - Hospital Universitario de Salamanca, Salamanca
  - Local Institution - 304, Salamanca
  - Hospital Universitario Virgen Del Rocio, Seville
  - Local Institution - 308, Seville
  - CEIC Hospital Universitario La Fe, Valencia
- United Kingdom (11):
  - Local Institution - 701, Boston
  - United Lincolnshire Hospitals NHS Trust, Boston
  - Cambridge University Hospitals NHS Foundation Trust, Addenbrooke's Hospital, Cambridge
  - Broomfield Hospital, Chelmsford
  - Saint James University Hospital, Leeds
  - King's College HospitalSchool of Medicine, London
  - Local Institution - 700, London
  - Hammersmith Hospital, London
  - University College London, London
  - Northwick Park Hospital, Middlesex
  - Southampton General Hospital, Southampton

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized at 33 sites globally. The sites were located in: Australia (3), Europe (18) and the United States (12).
Pre-assignment Details: Participants were eligible who did not respond to an adequate course of therapy with an injectable hypomethylating agent (iHMA - azacitidine or decitabine) or were unable to tolerate an iHMA following at least 3 months of attempted treatment.
Groups:
- Stable Disease (SD) Cohort: Oral Azacitidine: Participants were given oral azacitidine (AZA) 100 mg, 150 mg, or 200 mg tablets twice daily (BID) on days 1 to 21 of each 28-day treatment cycle. Participants continued to receive their assigned study treatment unless disease progression, unacceptable toxicity, lost to follow-up or withdrawal by participant occurred.
- Progressive Disease (PD) Cohort: Oral Azacitidine: Participants were given oral azacitidine 100 mg, 150mg, or 200mg tablets BID on days 1 to 21 of each 28-day treatment cycle. Participants continued to receive their assigned study treatment unless disease progression, unacceptable toxicity, lost to follow-up or withdrawal by participant occurred.
- Stable Disease Cohort: Oral Azacitidine and Durvalumab: Participants received 100 mg oral azacitidine (AZA) tablets BID on days 1 to 14 or days 1 to 21 of each 28-day treatment cycle and durvalumab (Durva) 1500 mg by intravenous infusion on day 1 of each 28-day treatment cycle; participants continued to receive their assigned study treatment unless disease progression, unacceptable toxicity, lost to follow-up or withdrawal by participant occurred.
- Progressive Disease Cohort: Oral Azacitidine and Durvalumab: Participants received 100 mg oral azacitidine tablets BID on days 1 to 14 or days 1 to 21 of each 28-day treatment cycle and durvalumab 1500 mg by intravenous infusion on day 1 of each 28-day treatment cycle; participants continued to receive their assigned study treatment unless disease progression, unacceptable toxicity, lost to follow-up or withdrawal by participant occurred.
Period: Overall Study
Arm/Group | Stable Disease (SD) Cohort: Oral Azacitidine | Progressive Disease (PD) Cohort: Oral Azacitidine | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab
Started | 32 | 22 | 6 | 5
Completed | 3 | 1 | 1 | 0
Not Completed | 29 | 21 | 5 | 5
Not completed — Death | 21 | 18 | 3 | 5
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 0
Not completed — Site Closure by Sponsor | 5 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat population included all enrolled participants who received at least one dose of investigational product (IP)..
Groups:
- Total: Total of all reporting groups
Arm/Group | Stable Disease (SD) Cohort: Oral Azacitidine | Progressive Disease (PD) Cohort: Oral Azacitidine | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab | Total
Number analyzed (Participants) | 32 | 22 | 6 | 5 | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.9 (7.62) | 75.1 (7.56) | 70.0 (7.21) | 72.4 (5.55) | 73.9 (7.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 0 | 0 | 19
  Male | 20 | 15 | 6 | 5 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 28 | 18 | 6 | 5 | 57
  Black | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Other | 1 | 1 | 0 | 0 | 2
  Not Collected or Reported | 2 | 0 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2 | 4
  Not Hispanic or Latino | 30 | 21 | 6 | 3 | 60
  Unknown | 1 | 0 | 0 | 0 | 1
Myelodysplastic Syndrome (MDS) World Health Organization Classification 2008 [Count of Participants; unit: Participants] — The World Health Organization (WHO) 2008 classification recognizes eight subtypes of MDS that are distinguished by the percentage of myeloblasts, presence or absence of ringed sideroblasts (i.e., erythroid precursors with iron deposits surrounding the nucleus), presence of a monocytosis or a deletion 5q.
  Participants
    Refractory Anemia (RA) with Ringed Sideroblasts | 1 | 0 | 0 | 0 | 1
    Refractory Cytopenia with Multilineage Dysplasia | 11 | 2 | 1 | 0 | 14
    RA With Excess Blasts-1 (RAEB-1) | 10 | 6 | 1 | 2 | 19
    RA With Excess Blasts-2 (RAEB-2) | 8 | 11 | 4 | 3 | 26
    MDS Unclassified (MDS-U) | 1 | 3 | 0 | 0 | 4
    MDS Associated with Isolated del (5q) | 0 | 0 | 0 | 0 | 0
    Missing | 1 | 0 | 0 | 0 | 1
International Prognostic Scoring System Risk Classification [Count of Participants; unit: Participants] — The international prognostic scoring system (IPSS) is a standard for risk assessment in primary myelodysplastic syndromes (MDS) that categorizes prognoses taking into account cytogenetics, cytopenias, blasts and blood counts. The IPSS prognostic subgroups consist of low-, intermediate-1-, intermediate-2-, and high-risk groups. The scale is 0-3.5 at 0.5 increments. Scores of 0=Low; 0.5-1.0=Int-1; 1.5-2.0=Int-2; 2.5-3.5=High risk which corresponds to poorer prognosis.
  Participants
    Low (0) | 4 | 2 | 0 | 0 | 6
    Intermediate 1 (0.5-1.0) | 12 | 5 | 1 | 2 | 20
    Intermediate (2) (1.0-2.0) | 7 | 7 | 4 | 2 | 20
    High (2) (≥ 2.5) | 8 | 8 | 1 | 1 | 18
    Unknown | 1 | 0 | 0 | 0 | 1
French-American-British (FAB) Classification [Count of Participants; unit: Participants] — FAB is a classification system for five (5) subtypes of myelodysplastic syndrome that are distinguished by the percentage of myeloblasts, presence or absence of ringed sideroblasts or a monocytosis.
  Participants
    Refractory Anemia (RA) | 6 | 2 | 0 | 0 | 8
    Refractory Anemia with Ringed Sideroblasts (RARS) | 6 | 1 | 1 | 0 | 8
    Refractory Anemia with Excess Blasts (RAEB) | 17 | 16 | 5 | 4 | 42
    RAEB in Transformation | 2 | 3 | 0 | 1 | 6
    Chronic Myelomonocytic Leukemia (CMML) | 0 | 0 | 0 | 0 | 0
    Missing | 1 | 0 | 0 | 0 | 1
Time Since Initial Diagnosis of MDS [Mean (Standard Deviation); unit: months] | 26.79 (29.678) | 26.97 (33.835) | 40.20 (61.663) | 23.51 (30.524) | 27.84 (34.266)
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — ECOG performance status is used by doctors and researchers to assess how a subject's disease is progressing, assess how the disease affects the daily living activities of the subject and determine appropriate treatment and prognosis. 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity)
  Participants
    0 (Fully active) | 5 | 6 | 3 | 2 | 16
    1 (Restricted but Ambulatory) | 22 | 13 | 3 | 3 | 41
    2 (Ambulatory But Unable to Work) | 5 | 3 | 0 | 0 | 8
    3 (Limited Self-Care) | 0 | 0 | 0 | 0 | 0
    4 (Completely Disabled) | 0 | 0 | 0 | 0 | 0
    5 (Death) | 0 | 0 | 0 | 0 | 0
Baseline Platelet Transfusion Status [Count of Participants; unit: Participants] — Baseline Platelet transfusion dependence is defined as ≥ 2 transfusions (in units) during the 56 days prior to treatment. Platelet transfusion independence is defined as 0 transfusions (in units) during the 56 days prior to treatment.
  Participants
    Dependent | 4 | 5 | 0 | 1 | 10
    Independent | 25 | 13 | 6 | 4 | 48
    Other | 3 | 4 | 0 | 0 | 7
Baseline Red Blood Cell (RBC) Transfusion Status [Count of Participants; unit: Participants] — Baseline RBC Transfusion Dependence is defined as ≥ 4 transfusions (in units) during the 56 days prior to treatment. RBC transfusion independence is defined as 0 transfusions (in units) during the 56 days prior to treatment.
  Participants
    Dependent | 8 | 7 | 0 | 2 | 17
    Independent | 8 | 6 | 3 | 2 | 19
    Other | 16 | 9 | 3 | 1 | 29
Average Red Blood Cell (RBC) Transfusion Requirement [Median (Full Range); unit: units per 56 days] — Documentation of all red blood cell transfusions received by the participant within 8 weeks (56 days) prior to the first dose of study drug.
  units per 56 days | 4.00 [0.00 to 10.0] | 3.50 [0.0 to 7.0] | 3.00 [0.0 to 7.0] | 4.00 [0.0 to 15.0] | 4.00 [0.0 to 15.0]

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate Based on the Modified International Working Group (IWG) 2006 Response Criteria for Myelodysplastic Syndrome (MDS)
Description: The overall response rate (ORR) was defined as the percentage of participants who achieved an objective response including: hematologic improvement (HI), partial remission (PR), complete remission (CR), or marrow complete remission (mCR). Hematologic response was defined as: • CR: ≤ 5% myeloblasts with normal maturation of all cell lines; peripheral blood (PB) shows: hemoglobin ≥11 g/dL, neutrophils ≥1.0x10^9/L, platelets ≥100x10^9/dL, blasts (0%) • PR: same as CR bone marrow (BM) shows blasts decreased by ≥ 50% over pre-treatment but still > 5%; cellularity and morphology not relevant • mCR: BM: ≤ 5% myeloblasts and decrease by ≥ 50% over pre-treatment PB, PB: if HI responses, noted in addition to mCR • HI: HI erythroid response (HI-E); HI neutrophil response (HI-N) ; HI platelet response (HI-P)
Time Frame: Response was assessed every 2 cycles following treatment during the first 6 cycles, then every 3 cycles thereafter; median duration of treatment = 5.26 and 3.81 months for SD/PD for oral AZA arms respectively, and 1.84 months for AZA and Durva SD/PD arms
Population: The intent-to-treat (ITT) population included all enrolled participants who received at least one dose of investigational product (IP).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Stable Disease (SD) Cohort: Oral Azacitidine | Progressive Disease (PD) Cohort: Oral Azacitidine | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab
Number analyzed (Participants) | 32 | 22 | 6 | 5
Percentage of Participants | 6.3 [0.8 to 20.8] | 4.5 [0.1 to 22.8] | 16.7 [0.4 to 64.1] | 0 [NA to NA] — Could not be estimated as there were 0 responders.

2. Secondary Outcome: Kaplan-Meier Estimate of Overall Survival
Description: Overall survival (OS) was defined as the time from randomization to death from any cause, and was calculated using date of first dose and date of death, or date of last follow-up for censored subjects.
Time Frame: From first dose till death due to any cause (Up to 91 months)
Population: The ITT population included all enrolled participants who received at least one dose of IP.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Stable Disease (SD) Cohort: Oral Azacitidine | Progressive Disease (PD) Cohort: Oral Azacitidine | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab
Number analyzed (Participants) | 32 | 22 | 6 | 5
Months | 17.00 [10.03 to 24.99] | 6.28 [4.50 to 15.19] | 14.70 [1.58 to NA] — Not calculated due to insufficient number of events | 14.56 [9.73 to NA] — Not calculated due to insufficient number of events

3. Secondary Outcome: Kaplan Meier Estimate of Time to Onset of First and Best Response
Description: Time to onset of first response was defined as the time between the date of first investigational product (IP) dose and the earliest date any response (CR, PR, mCR, or HI) was first observed. Participants who did not achieve any defined response during the treatment period were censored at the date of treatment discontinuation, disease progression, or death, whichever occurred first. Best response is the best recorded response or treatment outcome from the start of the study treatment until the end of the study treatment taking into account the requirements for confirmation of response.
Time Frame: as for outcome 1
Population: The ITT population included all enrolled participants who received at least one dose of IP.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Stable Disease (SD) Cohort: Oral Azacitidine | Progressive Disease (PD) Cohort: Oral Azacitidine | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab
Number analyzed (Participants) | 32 | 22 | 6 | 5
Months
  Onset of First Response | NA [10.85 to NA] — Could not be estimated due to the insufficient number of events. | 11.97 [NA to NA] — Could not be estimated due to the insufficient number of events. | NA [1.64 to NA] — Could not be estimated due to the insufficient number of events. | NA [NA to NA] — Could not be estimated due to the insufficient number of events.
  Onset of Best Response | 3.68 [2.10 to NA] — Could not be estimated due to the insufficient number of events. | 4.41 [1.68 to NA] — Could not be estimated due to the insufficient number of events. | 3.29 [1.64 to NA] — Could not be estimated due to the insufficient number of events. | 2.17 [1.64 to NA] — Could not be estimated due to the insufficient number of events.

4. Secondary Outcome: Kaplan Meier Estimate of Duration of First Response
Description: Duration of hematologic response and/or improvement was defined as the time from the date response or improvement was first observed to the date of documented relapse or disease progression as defined by the modified IWG 2006 criteria. Particpants who maintained hematologic response and/or improvement through the end of the treatment period were censored as the date of treatment discontinuation or death, whichever occurred first.
Time Frame: as for outcome 1
Population: The ITT population included all enrolled participants who received at least one dose of IP; participants who achieved a response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Stable Disease (SD) Cohort: Oral Azacitidine | Progressive Disease (PD) Cohort: Oral Azacitidine | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab
Number analyzed (Participants) | 3 | 2 | 1 | 0
Months | NA [9.24 to NA] — Could not be estimated due to the insufficient number of events. | NA [NA to NA] — Could not be estimated due to the insufficient number of events. | NA [NA to NA] — Could not be estimated due to the insufficient number of events. |

5. Secondary Outcome: Kaplan Meier Estimate of Duration of Best Response
Description: as for outcome 4
Time Frame: as for outcome 1
Population: The ITT population included all enrolled participants who received at least one dose of IP; participants who achieved a best response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Stable Disease (SD) Cohort: Oral Azacitidine | Progressive Disease (PD) Cohort: Oral Azacitidine | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab
Number analyzed (Participants) | 32 | 22 | 6 | 5
Months | NA [9.24 to NA] — Could not be estimated due to the insufficient number of events. | NA [NA to NA] — Could not be estimated due to the insufficient number of events. | NA [NA to NA] — Could not be estimated due to the insufficient number of events. | NA [NA to NA] — Could not be estimated due to the insufficient number of events.

6. Secondary Outcome: Kaplan-Meier Estimate of Progression Free Survival (PFS)
Description: Progression-free survival is defined as the time from first dose to the first documented progressive disease (PD), relapse, or death due to any cause during or after the treatment period, whichever occurred first, according to IWG 2006 response criteria for MDS. Participants who were still alive and progression-free were censored at the date of their last response assessment. Progressive disease is defined as follows: - an increase in BM blasts relative to nadir: •If nadir less than 5% blasts: ≥ 50% increase in blasts to > 5% blasts •If nadir 5% - 10% blasts: ≥ 50% increase in blasts to > 10% blasts •If nadir 10% - 20% blasts: ≥ 50% increase in blasts to > 20% blasts •If nadir 20% - 30% blasts: ≥ 50% increase in blasts to > 30% blasts And any of the following: •At least 50% decrement from maximum remission/response levels in granulocytes or platelets •Reduction in Hgb concentration by ≥ 2 g/dL •Transfusion dependence
Time Frame: From first dose to the first documented progressive disease (PD), relapse, or death due to any cause (Up to 91 months)
Population: The ITT population included all enrolled participants who received at least one dose of IP.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Stable Disease (SD) Cohort: Oral Azacitidine | Progressive Disease (PD) Cohort: Oral Azacitidine | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab
Number analyzed (Participants) | 32 | 22 | 6 | 5
Months | 14.86 [9.27 to 24.99] | 6.28 [4.50 to 15.19] | 14.70 [1.58 to NA] — Could not be estimated due to the insufficient number of events. | 12.10 [2.17 to NA] — Could not be estimated due to the insufficient number of events.

7. Secondary Outcome: Percentage of Participants With Progressive Disease at Baseline Who Achieved Stable Disease
Description: A participant was considered as having a stable disease if the disease neither responded nor progressed during or after study treatment.
Time Frame: as for outcome 1
Population: Includes participants who had progressive disease at baseline who achieved stable disease.
Measure: Number; unit: Percentage of Participants
Arm/Group | Stable Disease (SD) Cohort: Oral Azacitidine | Progressive Disease (PD) Cohort: Oral Azacitidine | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab
Number analyzed (Participants) | 0 | 22 | 0 | 5
Percentage of Participants |  | 36.4 |  | 20.0

8. Secondary Outcome: Kaplan-Meier Estimate of Onset to Achieve Stable Disease
Description: as for outcome 7
Time Frame: as for outcome 1
Population: Includes all participants in the ITT population with progressive disease at baseline and achieved stable disease; those who didn't achieve SD or better were censored.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Stable Disease (SD) Cohort: Oral Azacitidine | Progressive Disease (PD) Cohort: Oral Azacitidine | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab
Number analyzed (Participants) | 0 | 22 | 0 | 5
Months |  | NA [1.74 to NA] — Could not be estimated due to the insufficient number of events |  | NA [1.64 to NA] — Could not be estimated due to the insufficient number of events

9. Secondary Outcome: Kaplan-Meier Estimate of Duration of Stable Disease
Description: The duration of stable disease was defined as the time between any two observations of objective disease progression (modified IWG criteria), starting from the first day of dosing with IP. Participants who maintained stable disease through the end of the treatment period were censored at the date of study termination.
Time Frame: as for outcome 1
Population: The population includes participants who achieved stable disease as their best response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Stable Disease (SD) Cohort: Oral Azacitidine | Progressive Disease (PD) Cohort: Oral Azacitidine | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab
Number analyzed (Participants) | 32 | 22 | 0 | 5
Months | NA [10.85 to NA] — Could not be estimated due to the low number of events. | NA [10.16 to NA] — Could not be estimated due to the low number of events. |  | NA [NA to NA] — Could not be estimated due to the low number of events.

10. Secondary Outcome: Percentage of Participants Who Progressed to Acute Myelogenous Leukemia (AML)
Description: For all participants who received at least one dose of study drug, continuous monitoring for progression to AML occurred in the post treatment follow up period.
Time Frame: From first dose and until death, loss to follow-up, withdrawal of consent for further data collection (Up to 91 months)
Population: The ITT population included all enrolled participants who received at least one dose of IP.
Measure: Number; unit: Percentage of Participants
Arm/Group | Stable Disease (SD) Cohort: Oral Azacitidine | Progressive Disease (PD) Cohort: Oral Azacitidine | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab
Number analyzed (Participants) | 32 | 22 | 6 | 5
Percentage of Participants | 31.3 | 18.2 | 33.3 | 60.0

11. Secondary Outcome: Kaplan-Meier Estimate of Time to Progression to AML
Description: Time to AML progression was defined as the time from the date of first dose of IP until the date the participant had documented progression to AML.
Time Frame: From first dose and until death, loss to follow-up, withdrawal of consent for further data collection (Up to 91 months)
Population: The ITT population included all enrolled participants who received at least one dose of investigational product (IP).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Stable Disease (SD) Cohort: Oral Azacitidine | Progressive Disease (PD) Cohort: Oral Azacitidine | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab
Number analyzed (Participants) | 32 | 22 | 6 | 5
Months | NA [12.89 to NA] — Could not be estimated due to the insufficient number of events. | NA [8.42 to NA] — Could not be estimated due to the insufficient number of events. | 21.47 [1.68 to NA] — Could not be estimated due to the insufficient number of events. | 6.21 [1.64 to NA] — Could not be estimated due to the insufficient number of events.

12. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as AEs occurring or worsening on or after the date of the first dose of oral aza or durva and within 28 days after last dose of oral aza or 90 days after last dose of durva A serious adverse event (SAE) is any: • Death; • Life-threatening event; • Any inpatient hospitalization or prolongation of existing hospitalization; • Persistent or significant disability or incapacity; • Congenital anomaly or birth defect; • Any other important medical event The severity of an AE was evaluated by the investigator according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (Version 4.0) where Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening and Grade 5 = Death.
Time Frame: From first dose until 28 days after the last dose of CC-486 (90 days after the last dose of durvalumab) or the last follow up visit, whichever date is later (Up to 91 months)
Population: The safety population included all enrolled participants who received at least 1 dose of IP and had at least 1 post-dose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Stable Disease (SD) Cohort: Oral Azacitidine | Progressive Disease (PD) Cohort: Oral Azacitidine | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab
Number analyzed (Participants) | 32 | 22 | 6 | 5
Participants
  ≥ 1 TEAE | 32 | 22 | 6 | 5
  ≥ 1 TEAE Related to (R/T) Oral Azacitidine (AZA) | 28 | 20 | 6 | 4
  ≥ 1 TEAE R/T Durvalumab (Durva) | 0 | 0 | 5 | 4
  ≥ 1 TEAE R/T Oral AZA or Durva | 28 | 20 | 6 | 4
  ≥ 1 Serious TEAE | 25 | 15 | 4 | 5
  ≥ 1 Serious TEAE R/T Oral AZA | 4 | 3 | 2 | 1
  ≥ 1 Serious TEAE R/T Durva | 0 | 0 | 1 | 1
  ≥ 1 Serious TEAE R/T Oral AZA or Durva | 4 | 3 | 2 | 1
  ≥ 1 NCI CTC Grade (GR) 3 or 4 TEAE | 32 | 19 | 5 | 5
  ≥ 1 NCI CTC GR 3 or 4 TEAE R/T Oral AZA | 18 | 10 | 4 | 3
  ≥ 1 NCI CTC GR 3 or 4 TEAE R/T Durva | 0 | 0 | 2 | 2
  ≥ 1 NCI CTC GR 3 or 4 TEAE R/T AZA or Durva | 18 | 10 | 4 | 3
  ≥ 1 TEAE Leading to Death | 4 | 4 | 2 | 0
  ≥ 1 TEAE Leading to Death R/T Oral AZA | 0 | 0 | 0 | 0
  ≥ 1 TEAE Leading to Death R/T Durva | 0 | 0 | 0 | 0
  ≥ 1 TEAE Leading to Death R/T AZA or Durva | 0 | 0 | 0 | 0
  ≥ 1 TEAE Leading to Dose Reduction of AZA | 10 | 8 | 1 | 0
  ≥ 1 TEAE Leading to Reduction of Durva | 0 | 0 | 0 | 0
  ≥ 1 TEAE Leading to Reduction of AZA or Durva | 10 | 8 | 1 | 0
  ≥1 TEAE Leading to Interruption of AZA | 21 | 13 | 3 | 4
  ≥1 TEAE Leading to Interruption of Durva | 0 | 0 | 2 | 0
  ≥1 TEAE Leading to Interruption of AZA or Durva | 21 | 13 | 3 | 4
  ≥ 1 TEAE Leading to Discontinuation (D/C) of AZA | 15 | 8 | 4 | 4
  ≥ 1 TEAE Leading to D/C of Durva | 0 | 0 | 3 | 3
  ≥ 1 TEAE Leading to D/C of AZA or Durva | 15 | 8 | 4 | 4

13. Secondary Outcome: Serum Plasma Concentration of Azacitidine and Durvalumab
Description: Data was not collected
Time Frame: Day 1, 8, 15 and 22
Population: Pharmacokinetic population
Arm/Group | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Maximum Observed Concentration (Cmax) of Azacitidine and Durvalumab
Description: Data was not collected
Time Frame: Day 1, 8, 15 and 22
Population: Pharmacokinetic population
Arm/Group | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Area Under Curve (AUC) of Azacitidine and Durvalumab
Description: Data was not collected
Time Frame: Day 1, 8, 15 and 22
Population: Pharmacokinetic population
Arm/Group | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Time to Maximum Concentration (Tmax) of Azacitidine and Durvalumab
Description: Data was not collected
Time Frame: Day 1, 8, 15 and 22
Population: Pharmacokinetic population
Arm/Group | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Terminal Half-life ( ½) of Azacitidine and Durvalumab
Description: Data was not collected
Time Frame: Day 1, 8, 15 and 22
Population: Pharmacokinetic population
Arm/Group | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Clearance (CL/F) of Azacitidine and Durvalumab
Description: Data was not collected
Time Frame: Day 1, 8, 15 and 22
Population: Pharmacokinetic population
Arm/Group | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Volume of Distribution (Vz/F) of Azacitidine and Durvalumab
Description: Data was not collected
Time Frame: Day 1, 8, 15 and 22
Population: Pharmacokinetic population
Arm/Group | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: SAE and Non-SAEs were collected from first dose until 28 days after the last dose of CC-486 (90 days after the last dose of durvalumab) or the last follow up visit, whichever date is later (Up to 91 months). Participants were assessed for all-cause mortality from first dose till death due to any cause (Up to 91 months).
Description: The number at Risk for All-Cause Mortality represents all enrolled participants. The number at risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents safety population that include all enrolled subjects who have received at least 1 dose of IP and had at least 1 post-dose safety assessment.
Arm/Group | Stable Disease (SD) Cohort: Oral Azacitidine | Progressive Disease (PD) Cohort: Oral Azacitidine | Stable Disease Cohort: Oral Azacitidine and Durvalumab | Progressive Disease Cohort: Oral Azacitidine and Durvalumab
All-Cause Mortality (participants affected / at risk) | 22/32 | 18/22 | 3/6 | 5/5
Serious Adverse Events (participants affected / at risk) | 25/32 | 15/22 | 4/6 | 5/5
Other Adverse Events (participants affected / at risk) | 32/32 | 22/22 | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stable Disease (SD) Cohort: Oral Azacitidine (N=32) | Progressive Disease (PD) Cohort: Oral Azacitidine (N=22) | Stable Disease Cohort: Oral Azacitidine and Durvalumab (N=6) | Progressive Disease Cohort: Oral Azacitidine and Durvalumab (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 2 | 0
Hyperleukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 1 | 2
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis gangrenous (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Fungaemia (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 9 | 2 | 0 | 2
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 3 | 2 | 0 | 0
Serratia bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Transformation to acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 3 | 1 | 3
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0
Dementia (Nervous system disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stable Disease (SD) Cohort: Oral Azacitidine (N=32) | Progressive Disease (PD) Cohort: Oral Azacitidine (N=22) | Stable Disease Cohort: Oral Azacitidine and Durvalumab (N=6) | Progressive Disease Cohort: Oral Azacitidine and Durvalumab (N=5)
Anaemia (Blood and lymphatic system disorders) | 12 | 10 | 1 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 12 | 6 | 1 | 2
Splenomegaly (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 6 | 1 | 4
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 2
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 2
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Tricuspid valve disease (Cardiac disorders) | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 2 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1
Eye haemorrhage (Eye disorders) | 2 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Anal erythema (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 13 | 9 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 21 | 11 | 4 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 2 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 24 | 12 | 2 | 2
Oral mucosa haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 4 | 3 | 1 | 1
Vomiting (Gastrointestinal disorders) | 18 | 11 | 2 | 3
Asthenia (General disorders) | 9 | 4 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 1 | 0 | 1 | 1
Fatigue (General disorders) | 10 | 6 | 2 | 4
Generalised oedema (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 6 | 2 | 1 | 3
Pyrexia (General disorders) | 7 | 3 | 1 | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 2 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 3 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 5 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 2 | 0 | 2
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 2 | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 5 | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 0 | 0 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 4 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 3 | 1 | 0 | 0
Cardiac murmur (Investigations) | 1 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0
Serum ferritin increased (Investigations) | 2 | 0 | 0 | 0
Urine output decreased (Investigations) | 1 | 0 | 0 | 1
Weight decreased (Investigations) | 10 | 6 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 15 | 8 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0
Gout (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 1 | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 6 | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 4 | 1 | 1 | 0
Lethargy (Nervous system disorders) | 2 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 2 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 2 | 0 | 1
Insomnia (Psychiatric disorders) | 6 | 2 | 0 | 1
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 1 | 0 | 0
Renal cyst (Renal and urinary disorders) | 2 | 0 | 0 | 1
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 2 | 2 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 1 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 3
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT02281084/Prot_000.pdf
  • Statistical Analysis Plan (2015-09-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT02281084/SAP_001.pdf